CLINICAL TRIAL: NCT05754697
Title: Instrument Assisted Soft Tissue Mobilization Versus Positional Release Technique in Patients With Chronic Plantar Fasciitis
Brief Title: IASTM Versus PRT in Patients With Chronic PF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Said Mohamed Ibrahim, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003841
Record Dates: First submitted 2023-01-28; First posted 2023-03-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Plantar Fasciitis
Keywords: Positional release technique; Instrument assisted soft tissue mobilization
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- instrument assisted soft tissue mobilization in addition to traditional treatment (Experimental): study group
  Interventions: Other: Instrument assisted soft tissue mobilization in addition to traditional treatment
- positional release technique in addition to traditional treatment (Experimental): study group
  Interventions: Other: Positional release technique in addition to traditional treatment
- traditional treatment (Active Comparator): control group
  Interventions: Other: Traditional treatment

INTERVENTIONS:
Other: Instrument assisted soft tissue mobilization in addition to traditional treatment — The treatment protocol will be two sessions will be given per week for 4 weeks.
  Arms: instrument assisted soft tissue mobilization in addition to traditional treatment
Other: Positional release technique in addition to traditional treatment — The treatment protocol will be two sessions will be given per week for 4 weeks.
  Arms: positional release technique in addition to traditional treatment
Other: Traditional treatment — The treatment protocol will be two sessions will be given per week for 4 weeks.
  Arms: traditional treatment

SUMMARY:
The goal of this clinical trial] is to compare between the effect of instrument assisted soft tissue mobilization and positional release technique in patients with chronic plantar fasciitis

The main question[s] it aims to answer are:

1. Is there a difference between the effect of instrument assisted soft tissue mobilization and positional release technique on pain pressure threshold in patients with chronic plantar fasciitis?
2. Is there a difference between the effect of instrument assisted soft tissue mobilization and positional release technique on foot function level in patients with chronic plantar fasciitis?

DETAILED DESCRIPTION:
Design of the study:

Pretest - posttest randomized controlled trial.

Subjects selection:

Sixty patients their age range from 30-50 years of both genders with chronic plantar fasciitis will participate in this study according to sample size calculation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed cases of plantar fasciitis not less than 3 months.
2. Heel pain felt maximally over plantar aspect of heel.
3. Pain in the heel on the first step in the morning.
4. Their age ranging from 30-50 years.
5. Body mass index range from (18.5 to 24.9 kg/m2).

Exclusion Criteria:

1. Subjects can't tolerate close physical contact.
2. Athletes.
3. Subjects with skin infections.
4. Subjects with recent fracture with incomplete bony union.
5. Subjects with acute inflammatory or infectious process.
6. Subjects with hematoma.
7. Subjects with osteoporosis.
8. Subjects with foot deformity.
9. Subjects that take medications that may increase blood clotting.
10. Surgery to the ankle or foot.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Pressure Algometer (Change in pain pressure threshold) | Pre-intervention and immediately after intervention
  Change in pain pressure threshold as assessed using pressure algometer on medial plantar process, with the unit of measurement in kg/cm².
  Change in pain pressure threshold as assessed using pressure algometer on gastrocnemius muscle, with the unit of measurement in kg/cm².
  Change in pain pressure threshold as assessed using pressure algometer on soleus muscle, with the unit of measurement in kg/cm².
  Change in pain pressure threshold as assessed using pressure algometer over the posteromedial aspect of the calcaneus , with the unit of measurement in kg/cm².

SECONDARY OUTCOMES:
The Arabic Version of Foot and Ankle Ability Measure | Pre-intervention and immediately after intervention
  The foot and ankle ability measure is a reliable, responsive, and valid measure of physical function for individuals with a broad range of musculoskeletal disorders of the lower leg, foot, and ankle.
  This self-report outcome instrument is available in English, German, French and Persian. The Foot and Ankle Ability Measure is a 29-item questionnaire divided into two subscales: the Foot and Ankle Ability Measure, 21-item Activities of Daily Living Subscale and the Foot and Ankle Ability Measure, 8-item Sports Subscale.
  Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. Item score totals, which range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale, were transformed to percentage scores. Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Ibrahim, Principal Investigator — Cairo University
Locations (1):
- Private Clinic, Port Said, Egypt

IPD SHARING:
Plan to Share IPD: No